CLINICAL TRIAL: NCT01201226
Title: Can Dormant Ovarian Follicles From Perimenopausal Women Become Gonadotropin Responsive by Incubation With PTEN Inhibitor and PI3K Activating Peptide?
Brief Title: Can Dormant Perimenopausal Ovarian Follicles Become FSH Responsive?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Izhar Ben-Shlomo, MD, Senior Obstetrician & Gynecologist, Dept. Ob/Gyn, Baruch Padeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PrimordialFollicleActivat.CTIL
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Low Ovarian Reserve; Poor Responders to Gonadotropihins Treatment
Keywords: Primordial ovarian follicles; PTEN; PI3K activating peptide; Low ovarian reserve; Gonadotrophins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (No Intervention): Perimenopausal women, who will undergo oelvic organ surgery, and will allow harvest of about half an oary for the study purpose
  Interventions: Other: Removal of half an ovary

INTERVENTIONS:
Other: Removal of half an ovary — Removal of half an ovary

SUMMARY:
The purpose of this study to obtain ovarian cortical fragments from perimenopausal patients, who undergo pelvic organ surgery and test whether treatment with PTEN inhibitor and PI3K activating peptide would induce these fragments to produce FSH responsive follicles in the nude mouse model.

DETAILED DESCRIPTION:
Introduction Women stop menstruating at the mean age of 51, yet pregnancies become much less prevalent beyond 40, with pregnancy at 43 being a relative rarity. Current common perception attributes the regression of fertility to depletion of the primordial follicles' pool (Burger et al. 2008). The decline in fertility may result not necessarily from a sharp depletion of the primordial follicle pool (Hansen et al. 2008) but may be due to failure of adequate transition from primordial to antral, gonadotropin-responsive follicles. It is not infrequent to encounter a fertility patient at her late thirties or early forties, who would not respond to the most extreme doses of exogenous FSH, but will nevertheless continue to menstruate until the age of 50. The usual practice is to refer these patients to oocyte donation programs.

Recently, Li et al. (2010) demonstrated that incubation of neonatal mouse ovarian fragments with an inhibitor of the Phosphatase with TENsin homology deleted in chromosome 10 (PTEN) phosphatase and a PI3K activating peptide, increased nuclear exclusion of Foxo3 and propelled large numbers of dormant primordial follicles into becoming FSH-responsive antral follicles. Furthermore, in the nude mice model (mice lacking immune system) they showed that transplanted human ovarian fragments containing mainly primordial follicles from surgical specimens, treated by the same incubation, also underwent activation of dormant follicles to derive preovulatory follicles containing mature oocytes.

Based on all the above we hypothesize, that ovaries of women at their perimenopausal years could be propelled to become FSH-responsive, using incubation with PTEN inhibitor and PI3K activating peptide to activate dormant primordial follicles.

If found feasible, this technique could provide hope of achieving fertility to patients who would otherwise be referred to receive oocyte donation.

Aim of the proposed study To obtain ovarian cortical fragments from perimenopausal patients, who undergo gynecological surgery, and test whether treatment with PTEN phosphatase and PI3K activating peptide would induce these fragments to produce FSH responsive follicles in the nude mouse model.

Study subjects and specimen harvest Up to ten women, older than 45 years, who are scheduled to gynecological operation, will be asked to provide half of an ovary for the study. The tissue will then be cut to multiple fragments, suitable for cryopreservation.

Laboratory methods Cryopreservation of ovarian fragments will use a vitrification protocol similar to earlier report for oocyte cryo-storage (Yoon et al. 2003). Because the cryo-preservation reagents can easily penetrate primordial follicles as compared with the large oocytes, we anticipate efficient preservation of these follicles. In young patients, one 1 mm cortical cubes contains ~50 primordial follicles.

Three tissue samples from each patient will be transferred to the Hsueh laboratory in Stanford (attached letter), and will be thawed for in vitro activation followed by xeno-transplantation using the same protocol as that described by Li et al. from that laboratory. (Li et al. 2010). The in vitro incubation will be in bpV(pic) (Calbiochem), a PTEN inhibitor, which allows the activation of dormant follicles. and a cell-permeable phospho-peptide (740Y-P) (Tocris) capable of binding to the SH2 domain of the p85 regulatory subunit of PI3K to stimulate enzyme activity. Activated PI3K converts phosphatidylinositol (4, 5)-bisphosphate (PIP2) to phosphatidylinositol (3-5)-trisphosphate (PIP3), whereas the PTEN inhibitor prevents the conversion of PIP3 back to PIP2. Accumulated PIP3, in turn, could stimulate the phosphorylation of Akt and increase the nuclear exclusion of the transcriptional factor Foxo3.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 45 years, undergoing pelvic organ surgery

Exclusion Criteria:

* None

Ages: 45 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Ability of primordial follicles to respond to FSH after incubation | Two weeks
  Human ovarian fragments will be incubated with PTEN inhibitor and PI3K activating peptide and will then be transplanted to nude mice. Subsequently mice will recieve FSH, and follicular response will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Izhar Ben-Shlomo, MD, Study Chair — Dept. Ob/Gyn, Baruch Padeh Medical Center, Poria, Israel
Locations (1):
- Department of Obstetrics and Gynecology, Baruch Padeh Medical Center, Poria, Tiberias, Israel

REFERENCES:
- [Result] Hansen KR, Knowlton NS, Thyer AC, Charleston JS, Soules MR, Klein NA. A new model of reproductive aging: the decline in ovarian non-growing follicle number from birth to menopause. Hum Reprod. 2008 Mar;23(3):699-708. doi: 10.1093/humrep/dem408. Epub 2008 Jan 11. PMID 18192670
- [Result] Li J, Kawamura K, Cheng Y, Liu S, Klein C, Liu S, Duan EK, Hsueh AJ. Activation of dormant ovarian follicles to generate mature eggs. Proc Natl Acad Sci U S A. 2010 Jun 1;107(22):10280-4. doi: 10.1073/pnas.1001198107. Epub 2010 May 17. PMID 20479243
- [Result] Yoon TK, Kim TJ, Park SE, Hong SW, Ko JJ, Chung HM, Cha KY. Live births after vitrification of oocytes in a stimulated in vitro fertilization-embryo transfer program. Fertil Steril. 2003 Jun;79(6):1323-6. doi: 10.1016/s0015-0282(03)00258-9. PMID 12798878